CLINICAL TRIAL: NCT01231906
Title: A Phase III Randomized Trial of Adding Vincristine-Topotecan-Cyclophosphamide to Standard Chemotherapy in Initial Treatment of Non-Metastatic Ewing Sarcoma
Brief Title: Combination Chemotherapy in Treating Patients With Non-Metastatic Extracranial Ewing Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEWS1031; NCI-2011-02611 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S12-01231; CDR0000687639; COG-AEWS1031; AEWS1031 (Other: Children's Oncology Group); AEWS1031 (Other: CTEP); P30CA013330 (NIH); U10CA098543 (NIH); U10CA180830 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Localized Extraskeletal Ewing Sarcoma; Peripheral Primitive Neuroectodermal Tumor of Bone; Peripheral Primitive Neuroectodermal Tumor of Soft Tissues
MeSH Terms: interventions — Cyclophosphamide; Dexrazoxane; Razoxane; Doxorubicin; Etoposide; Ifosfamide; Topotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (combination chemotherapy) (Experimental): INDUCTION THERAPY: Patients receive vincristine sulfate IV on day 1 in weeks 1, 2, 5, 6, 9, and 10; doxorubicin hydrochloride IV over 1-15 minutes (or as per institutional policies up to 60-minutes) on days 1 and 2 and cyclophosphamide IV over 30-60 minutes on day 1 in weeks 1, 5, and 9; and ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 in weeks 3, 7, and 11.
  CONSOLIDATION THERAPY: Patients receive vincristine sulfate IV on day 1 in weeks 1, 2, 7, 8, 9, 10, 13, 14, 17, 18, 21, and 22; doxorubicin hydrochloride IV on days 1 and 2 in weeks 1 and 9; cyclophosphamide IV over 30-60 minutes on day 1 in weeks 1, 7, 9, 13, 17, and 21; and ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 in weeks 3, 5, 11, 15, and 19. Patients received Dexrazoxane with doxorubicin hydrochloride in weeks 1 and 9.
  Interventions: Drug: Cyclophosphamide; Drug: Dexrazoxane; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Vincristine Sulfate
- Arm B (combination chemotherapy, topotecan hydrochloride) (Experimental): INDUCTION THERAPY: Patients receive vincristine sulfate IV on day 1 in weeks 1, 2, 5, 6, 9, 10, 11 and 12; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1 and 9; cyclophosphamide IV over 15-30 minutes on days 1-5 in weeks 1 and 9, and over 30-60 minutes on day 1 of weeks 5 and 11; ifosfamide and etoposide as in arm A; and doxorubicin hydrochloride IV on days 1 and 2 in weeks 5 and 11.
  CONSOLIDATION THERAPY: Patients receive vincristine sulfate IV on day 1 in weeks 1, 2, 7-10, 13-16, 19, and 20; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1, 7, and 15; cyclophosphamide IV over 15-60 minutes on days 1-5 in weeks 1, 7, and 15, and over 30-60 minutes on day 1 in weeks 9, 13, and 19; ifosfamide IV over 1 hour and etoposide IV over 1- 2 hours on days 1-5 in weeks 3, 5, 11, 17, and 21; and doxorubicin hydrochloride IV on days 1 and 2 in weeks 9,13, and 19. Patients received Dexrazoxane with doxorubicin hydrochloride in weeks 13 and 19.
  Interventions: Drug: Cyclophosphamide; Drug: Dexrazoxane; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Dexrazoxane
  Other Names: 2, 6-Piperazinedione, 4,4'-propylenedi-, (P)- (8CI); 2,6-Piperazinedione, 4, 4'-(1-methyl-1,2-ethanediyl)bis-, (S)- (9CI); ADR 529; ADR-529; ADR529; ICRF 187; ICRF-187; ICRF187; Razoxane (+)-form; Soluble ICRF (L-isomer)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm B (combination chemotherapy, topotecan hydrochloride)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This trial examined the outcome benefit to patients of adding a new chemotherapy drug combination to the established treatment approach for patients with extracranial Ewing sarcoma, that had not spread from the primary site to other places in the body. The trial randomly assigned patients at the time of study entry to receive established standard treatment with the following 5-drugs: vincristine sulfate, doxorubicin hydrochloride, cyclophosphamide, ifosfamide and etoposide. The outcome for patients receiving the standard 5-drug combination was compared to the outcome for patients who received the same 5-drugs with an additional drug, topotecan hydrochloride delivered in a novel combination with vincristine sulfate and cyclophosphamide.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. Test the effect of the combination of vincristine (vincristine sulfate), cyclophosphamide, and topotecan (topotecan hydrochloride) (VTC) added to the standard 5-drug interval-compressed chemotherapy backbone on event-free and overall survival of children and young adults with Ewing sarcoma.

CORRELATIVE SCIENCE OBJECTIVES:

I. To evaluate initial volumetric tumor size as a prognostic factor for event free survival (EFS) in patients with localized Ewing tumors.

II. To evaluate histologic response as a prognostic factor for EFS in patients with localized Ewing tumors.

III. To continue evaluation of biologic markers both as related to prognosis and as eventual therapeutic targets via encouraging concurrent enrollment on a Ewing sarcoma specimen-collection study.

IV. To evaluate imaging response by fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) as a prognostic factor for EFS.

V. To evaluate the effects of the type of local therapy on EFS and overall survival.

VI. To evaluate the effect of local surgical margins in conjunction with histologic response on EFS in patients with localized Ewing tumors.

VII. To evaluate the effect of local therapy modality (surgery, radiotherapy, or a combination) as well as the type of surgical reconstruction on musculoskeletal complications.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A:

INDUCTION THERAPY: Patients receive vincristine sulfate intravenously (IV) on day 1 in weeks 1, 2, 5, 6, 9, and 10; doxorubicin hydrochloride IV over 1-15 minutes (or as per institutional policies up to 60-minutes) on days 1 and 2 and cyclophosphamide IV over 30-60 minutes on day 1 in weeks 1, 5, and 9; and ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 in weeks 3, 7, and 11.

CONSOLIDATION THERAPY: Patients receive vincristine sulfate IV on day 1 in weeks 1, 2, 7, 8, 9, 10, 13, 14, 17, 18, 21, and 22; doxorubicin hydrochloride IV on days 1 and 2 in weeks 1 and 9; cyclophosphamide IV over 30-60 minutes on day 1 in weeks 1, 7, 9, 13, 17, and 21; and ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 in weeks 3, 5, 11, 15, and 19. Patients received Dexrazoxane with doxorubicin hydrochloride in weeks 1 and 9.

ARM B:

INDUCTION THERAPY: Patients receive vincristine sulfate IV on day 1 in weeks 1, 2, 5, 6, 9, 10, 11 and 12; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1 and 9; cyclophosphamide IV over 15-30 minutes on days 1-5 in weeks 1 and 9, and over 30-60 minutes on day 1 of weeks 5 and 11; ifosfamide and etoposide as in arm A; and doxorubicin hydrochloride IV on days 1 and 2 in weeks 5 and 11.

CONSOLIDATION THERAPY: Patients receive vincristine sulfate IV on day 1 in weeks 1, 2, 7-10, 13-16, 19, and 20; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1, 7, and 15; cyclophosphamide IV over 15-60 minutes on days 1-5 in weeks 1, 7, and 15, and over 30-60 minutes on day 1 in weeks 9, 13, and 19; ifosfamide IV over 1 hour and etoposide IV over 1- 2 hours on days 1-5 in weeks 3, 5, 11, 17, and 21; and doxorubicin hydrochloride IV on days 1 and 2 in weeks 9,13, and 19. Patients received Dexrazoxane with doxorubicin hydrochloride in weeks 13 and 19.

Patients could undergo surgery alone after recovery from week 12 chemotherapy if the primary tumor could be completely resected with negative margins and with reasonable functional result. Patients with inadequate margins after surgery were to receive radiotherapy in addition. Patients with lesions in surgically difficult sites such as the spine, skull, and periacetabular pelvis, patients with a poor response to induction chemotherapy, or those patients in whom surgery would result in unacceptable functional results were recommended to receive radiation and not surgery. Radiotherapy was to be administered during weeks 1-7 of consolidation therapy or after recovery from surgery for patients with positive margins. Patients who received planned pre-operative radiation and had positive surgical margins were to receive additional radiotherapy.

After completion of study therapy, patients are followed up every 3 months for 3 years and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, biopsy confirmed, extracranial, non-metastatic Ewing sarcoma or primitive neuroectodermal tumor (PNET) of bone or soft tissue are eligible for this study; note:

  * For the purpose of this study, chest wall tumors with ipsilateral pleural effusions, ipsilateral positive pleural fluid cytology or ipsilateral pleural based secondary tumor nodules will be considered localized disease
  * Patients with regional node involvement, based on clinical suspicion confirmed by pathologic documentation are considered to be non-metastatic
  * Patients with discontinuous osseous lesions within the same bone are considered to be non-metastatic
  * Tumors arising in the bony skull (extra-dural) are considered to be extracranial
* Patient eligibility will be based on a diagnosis of Ewing sarcoma or PNET by institutional pathologist
* No prior chemotherapy or radiation therapy is allowed; patients should only have had a biopsy of the primary tumor without an attempt at complete or partial resection; patients will still be eligible if unplanned excision was attempted or accomplished as long as adequate imaging was obtained prior to surgery
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70mL/min/1.73 m^2 or serum creatinine based on age/gender as follows:

  * 1 month to < 6 months: 0.4 mg/dL
  * 6 months to < 1 year: 0.5 mg/dL
  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mg/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 13 to < 16 years: 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male), 1.4 mg/dL (female)
* Total bilirubin < 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN) for age
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by radionuclide angiogram

Exclusion Criteria:

* Patients must have no evidence of metastatic disease; metastatic disease are lesions which are discontinuous from the primary tumor, are not regional lymph nodes and do not share a body cavity with the primary tumor; if there is any doubt whether lesions are metastatic, a biopsy of those lesions should be taken

  * Skeletal lesions in adjacent bones (trans-articular)
  * Contralateral pleural effusion and contralateral pleural nodules
  * Distant lymph node involvement
  * Patients with pulmonary nodules are considered to have metastatic disease if the patient has:

    * Solitary nodule > 0.5 cm or multiple nodules of > 0.3 cm unless biopsied and negative for Ewing's
    * Biopsies of solitary nodule =< 0.5 cm or multiple nodules =< 0.3 cm are not required but if performed and positive indicate metastatic disease
* Patients whose tumors arise in the dural and intra-dural soft tissues of the cranium and spine are not eligible
* Patients with pathologic diagnoses other than Ewing sarcoma will be excluded
* Patients diagnosed with Ewing Sarcoma as a second malignant neoplasm are not eligible if they have received chemotherapy or radiation for the treatment of their primary malignancy
* Pregnant women will not be entered on this study; pregnancy tests must be obtained in female patients who are post-menarchal; lactating females may not participate unless they have agreed not to breastfeed their infants; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of the study treatment
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 642 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Leavey, Principal Investigator — Children's Oncology Group
Locations (243):
- United States (215):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Leavey PJ, Laack NN, Krailo MD, Buxton A, Randall RL, DuBois SG, Reed DR, Grier HE, Hawkins DS, Pawel B, Nadel H, Womer RB, Letson GD, Bernstein M, Brown K, Maciej A, Chuba P, Ahmed AA, Indelicato DJ, Wang D, Marina N, Gorlick R, Janeway KA, Mascarenhas L. Phase III Trial Adding Vincristine-Topotecan-Cyclophosphamide to the Initial Treatment of Patients With Nonmetastatic Ewing Sarcoma: A Children's Oncology Group Report. J Clin Oncol. 2021 Dec 20;39(36):4029-4038. doi: 10.1200/JCO.21.00358. Epub 2021 Oct 15. PMID 34652968
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy, Topotecan Hydrochloride)
Started (Eligible and began receiving protocol therapy) | 319 | 323
Received Therapy | 308 | 318
Completed (Completion of planned therapy with no event observed: disease progression, second malignant neoplasm (SMN), death regardless of cause) | 198 | 222
Not Completed | 121 | 101
Not completed — Lack of Efficacy | 75 | 68
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 34 | 24
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Ineligible | 10 | 3
Not completed — No treatment | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy, Topotecan Hydrochloride) | Total
Number analyzed (Participants) | 319 | 323 | 642
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 272 | 280 | 552
  Between 18 and 65 years | 47 | 43 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 13 [0 to 32] | 13 [0 to 34] | 13 [0 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 130 | 275
  Male | 174 | 193 | 367
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 44 | 89
  Not Hispanic or Latino | 269 | 275 | 544
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 11 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 10 | 4 | 14
  White | 267 | 280 | 547
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 28 | 56
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 286 | 286 | 572
  Australia | 17 | 20 | 37
  Canada | 14 | 13 | 27
  New Zealand | 2 | 2 | 4
  Saudi Arabia | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival
Description: Estimated 5-year EFS where EFS is calculated as the time from study enrollment to disease progression, disease relapse, occurrence of a second malignant neoplasm, death from any cause or last follow-up whichever occurs first. Kaplan-Meier method is used for estimation. Patients without an event are censored at last contact.
Time Frame: 5 years after enrollment
Population: Only eligible patients are considered in the calculation of this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy, Topotecan Hydrochloride)
Number analyzed (Participants) | 309 | 320
Percent Probability | 77.64 [72.42 to 81.99] | 78.79 [73.70 to 83.01]

2. Other Pre Specified Outcome: Overall Survival
Description: Time from study enrollment to death or last patient contact.
Time Frame: 5 years after enrollment
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Histological Response, in Terms of Event Free Survival After Local Control in Patients Who Received Local Control Therapy
Description: Percent of viable tumor in the resected tumor specimen after the patient receives 2 cycles of induction chemotherapy. Patients will be classified into groups according to: (1) good risk - less than 10% viable tumor in the resection specimen; and (2) standard risk - 10% or more viable tumor in the resection specimen. Patients who receive radiation therapy to the primary tumor prior to tumor resection or whose tumor is resected prior to the start of systemic therapy are not evaluable for this outcome measure.
Time Frame: At the end of INDUCTION THERAPY (84 days)
Reporting Status: Not Posted

4. Other Pre Specified Outcome: SUVmax as Determined by Positron Emission Tomography (PET)-Determined Response at Enrollment
Description: Patients will be classified into two groups according to SUVmax as: (1) study population median or greater; and (2) less than the study population median.
Time Frame: At study enrollment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: SUVmax as Determined by Positron Emission Tomography (PET)-Determined Response After Induction
Description: Patients will be classified into two groups according to SUVmax as: (1) study population median or greater; and (2) less than the study population median. Patients who receive radiation therapy to the primary tumor prior to the completion of 2 cycles of induction or who do not receive 2 cycles of induction chemotherapy are not evaluable for this outcome measure.
Time Frame: At the end of INDUCTION THERAPY (84 days)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Tumor Volume in Milliliters (ml) at Enrollment
Description: Patients will be classified into two groups: (1) tumor volume 200 ml or greater and (2) tumor volume less than 200 ml.
Time Frame: At study enrollment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Radiological Response of Soft Tissue Component of Mass by Radiological Evaluation at the End of Induction Chemotherapy
Description: Patients will be classified into two groups: (1) complete resolution of soft tissue mass; and (2) soft tissue mass present after induction chemotherapy. Patients who receive radiation therapy to the primary tumor prior to the completion of 2 cycles of induction, who do not receive 2 cycles of induction chemotherapy or who do not have soft tissue involvement detected at enrollment or at any time prior to the end of induction chemotherapy are not evaluable for this outcome measure.
Time Frame: At the end of INDUCTION THERAPY (84 days)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Type of Local Control Modality Used for Removal of Primary Tumor Site at Any Time up to the End of the First 6 Cycles of Consolidation Chemotherapy
Description: Patients will be categorized into the following groups: (1) surgery as the local control modality; (2) radiation therapy as the local control modality; (3) surgery and radiation therapy as the local control modality; and (4) no local control modality administered to the primary tumor site. Patients who do not complete induction chemotherapy will not be evaluable for this outcome measure.
Time Frame: 126 days after enrollment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Occurrence of Grade 2 or Higher Musculoskeletal Event (ME), or Surgery Required to Treat a Complication of Local Therapy
Description: Any National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 ME of grade 2 or greater or ME of any grade where surgery is required to treat a complication of local therapy. Patients who do not complete induction chemotherapy or do not have any local control modality administered to the primary tumor site will not be evaluable for this outcome measure.
Time Frame: 132 days after enrollment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Presence of Tumor at the Margin of Resection for Patients Who Have Surgery as the Only Local Control Modality
Description: Patients will be categorized into the following groups: (1) tumor present at the margin of resection; and (2) no tumor present at the margin of resection. Patients who are not classified as having surgery as the only local control modality will not be evaluable for this outcome measure.
Time Frame: 126 days after enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 months post-treatment planned as 252 days; All-Cause Mortality: up to 9 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy, Topotecan Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 51/308 | 42/318
Serious Adverse Events (participants affected / at risk) | 8/308 | 11/318
Other Adverse Events (participants affected / at risk) | 105/308 | 91/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Combination Chemotherapy) (N=308) | Arm B (Combination Chemotherapy, Topotecan Hydrochloride) (N=318)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Combination Chemotherapy) (N=308) | Arm B (Combination Chemotherapy, Topotecan Hydrochloride) (N=318)
Anemia (Blood and lymphatic system disorders) | 16 (16) | 16 (16)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 (28) | 25 (25)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cecal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 14 (14) | 7 (7)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fever (General disorders) | 3 (3) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (5) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 15 (15) | 6 (6)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 3 (3)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Soft tissue infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 4 (4) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (5) | 4 (4)
Neutrophil count decreased (Investigations) | 26 (26) | 26 (26)
Platelet count decreased (Investigations) | 23 (23) | 22 (22)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 17 (17) | 13 (13)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 13 (13)
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 5 (5)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT01231906/Prot_SAP_000.pdf